CLINICAL TRIAL: NCT05848713
Title: AntiThrombotic Therapy to Ameliorate Clinical Complications in Community Acquired Pneumonia
Acronym: ATTACC-CAP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Research Manitoba (Other); Ozmosis Research Inc. (Industry); Canadian Venous Thromboembolism Clinical Trials and Outcomes Research (CanVECTOR) Network (Network); Canadian Critical Care Trials Group (Other); AVANTI (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATTACC-CAP; OZM-129 (Other: Ozmosis Research Inc.)
Record Dates: First submitted 2023-04-17; First posted 2023-05-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Community-acquired Pneumonia
Keywords: Pneumonia; Heparin; Anticoagulation; Community acquired pneumonia; Unfractionated Heparin; Low Molecular Weight Heparin; Dalteparin; Enoxaparin; Tinzaparin
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia | interventions — Heparin

STUDY DESIGN:
Intervention Model Description: Adaptive stratified randomized clinical trial with Bayesian stopping rules
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapeutic-Dose Heparin (Experimental): Participants randomized to the investigational arm will receive a pragmatic strategy of therapeutic-dose low molecular-weight heparin (LMWH) or unfractionated heparin (UFH) administered daily for up to 14 days or until hospital discharge, whichever occurs first. Participants should start receiving study drug as soon as possible following randomization.
  Interventions: Drug: Heparin
- Usual Care (No Intervention): Participants randomized to the control arm will receive usual care thromboprophylactic dose anticoagulation according to local practice. To ensure adequate separation between the study groups, the dose of heparin/LMWH used in the usual care arm should not equal more than half of the approved therapeutic dose for that agent according to local VTE treatment protocols.

INTERVENTIONS:
Drug: Heparin — Preference is for LMWH given ease of administration and possibility of a more favorable safety profile, if no contraindication is present. Enoxaparin, dalteparin, or tinzaparin are acceptable LMWHs to be used for patients in the investigational arm and dose should be based on measured or estimated weight of the patient.
  Alternatively, intravenous UFH may be used and may be preferred in the presence of significant renal compromise. Intravenous UFH is typically dosed according to total body weight and pragmatically adjusted according to local institutional policy to achieve an activated partial thromboplastin time (aPTT) of 1.5-2.5x the reference value, or a corresponding UFH anti-Xa level. If UFH is used, the availability of a local site policy that specifies an aPTT target in this range or a corresponding anti-Xa value is a requirement.
  Arms: Therapeutic-Dose Heparin

SUMMARY:
This is an international, open-label, stratified randomized controlled trial with Bayesian adaptive stopping rules to compare the effects of therapeutic-dose heparin vs. usual care pharmacological thromboprophylaxis on outcomes in patients admitted to hospital with community acquired pneumonia (CAP).

DETAILED DESCRIPTION:
The global incidence of hospitalization due to CAP is high and associated with substantive morbidity and mortality. Thrombotic complications - including venous, arterial, and possibly microvascular - occur commonly in hospitalized patients across many etiologies of CAP. Poor outcomes may be mediated by both inflammatory and thrombotic processes leading to respiratory, cardiac, and other end organ dysfunction. There are currently no established therapies that modify the potentially maladaptive immunothrombosis pathway in CAP.

Therapeutic-dose anticoagulation with heparin reduces disease progression and mortality in non-critically ill patients hospitalized with COVID-19 with an acceptable safety profile. COVID-19 shares pathogenic features, including activation of the inflammatory and coagulation cascades, with other pneumonias. Whether therapeutic-dose heparin confers similar clinical benefits in non-COVID-19 CAP is unknown.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years of age
2. Admitted to hospital for a suspected or confirmed diagnosis of CAP defined by:

   1. Radiographic evidence of new or worsening infiltrate
   2. One or more of the following signs and/or symptoms of lower respiratory tract infection

   i. New or increased cough or sputum production ii. Fever of > 37.8C or temperature < 36C iii. WBC > 11 x 109/L or < 4 x 109/L c. The primary diagnosis is believed to be CAP as per the attending physician
3. Requires supplemental oxygen to treat hypoxemia (or requires an increased level of supplemental oxygen if on chronic oxygen therapy)
4. Hospital admission anticipated to last ≥72 hours from randomization

Exclusion Criteria:

1. Suspected or confirmed active COVID-19 infection
2. Hospital admission for >72 hours prior to randomization
3. Patients receiving non-invasive or invasive ventilation, vasopressors, or extracorporeal life support (ECLS) within an ICU at the time of enrollment
4. Requirement for chronic mechanical ventilation via tracheostomy prior to hospitalization
5. Patients for whom the intent is to not use pharmacologic thromboprophylaxis
6. Patients with an independent indication for therapeutic-dose anticoagulation
7. Patients with a contraindication to therapeutic-dose anticoagulation, including:

   1. Non-traumatic bleeding that requires medical evaluation or hospitalization within 30 days prior to CAP hospital admission
   2. History of an inherited or acquired bleeding disorder
   3. Cerebral aneurysm or mass lesions of the central nervous system
   4. Ischemic stroke within 3 months of hospital admission
   5. Gastrointestinal bleeding within 3 months of hospital admission
   6. Platelet count <50 x109/L OR INR >2.0 OR hemoglobin <80 g/L at the time of screening
   7. Other physician-perceived contraindications to therapeutic anticoagulation
8. History of heparin induced thrombocytopenia (HIT) or other heparin allergy
9. Current or recent (within 7 days of screening) use of dual anti-platelet inhibitors (For example; Aspirin + one of the following; clopidogrel, ticagrelor, prasugrel)
10. Patients in whom imminent death is anticipated
11. Anticipated transfer to another hospital that is not a study site within 72 hours of randomization
12. Enrollment in other interventional trials related to anticoagulation or antiplatelet therapy during current hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Ordinal endpoint reflecting survival | 30 days
  Survival to hospital discharge without ICU-level organ support. Organ support is defined as receipt of high flow nasal oxygen, invasive or non-invasive mechanical ventilation, vasopressor/inotropic therapy, or extracorporeal life support (ECLS) within an ICU. This outcome reflects disease progression to ICU-level organ failure or the worst possible outcome (death). It was chosen because of its importance to patients, clinicians, and other stakeholders. Given the limited number of ICU beds, reducing the burden of critical illness has important health system capacity implications.

SECONDARY OUTCOMES:
Bleeding events | 14 days
  Number of participants with major bleeds as defined by the ISTH definition.
HIT events | 14 days
  Number of participants with laboratory confirmed heparin induced thrombocytopenia (HIT)
Thrombotic events | 30 days and 90 days
  Number of participants with deep vein thrombosis, pulmonary embolism, systemic arterial thromboembolism, myocardial infarction, or ischemic stroke
Invasive mechanical ventilation | 30 days
  Ordered categorical endpoint with three possible outcomes based on the worst status of each patient through day 30 following randomization
All cause mortality | 30 days, 90 days, and 180 days
Hospital-free days | 30 days, 90 days, and 180 days
  Days alive outside hospital
Health related quality of life | 30 days, 90 days, and 180 days
  Using the EQ-5D-5L instrument
Health related quality of life | 30 days, 90 days, and 180 days
  Using the Clinical Frailty Scale instrument

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Zarychanski, MD, Principal Investigator — University of Manitoba; Patrick Lawler, MD, Principal Investigator — University Health Network and McGill University; Sylvain Lother, MD, Principal Investigator — University of Manitoba; Alexis Turgeon, MD, Principal Investigator — L'Universite Laval
Locations (62):
- United States (6):
  - University of Chicago, Chicago, Illinois
  - Ochsner Clinic, Jefferson, Louisiana
  - Maine Medical Centre, Portland, Maine
  - Henry Ford Health System, Dearborn, Michigan
  - Cooper University Health Care, Camden, New Jersey
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Brazil (31):
  - Hospital Estadual Dr. Jayme Santos Neves, Serra, Espírito Santo
  - Hospital Evangelico de Vila Velha, Vila Velha, Espírito Santo
  - Hospital Universitário Cassiano Antonio Moraes, Vitória, Espírito Santo
  - Santa Casa de Misericordia de Itabuna, Itabuna, Estado de Bahia
  - Hospital Brasilia, Brasília, Federal District
  - Hospital Sao Brasilia, Brasília, Federal District
  - Instituto de Cardiologia e Transplantes do Distrito Federal, Brasília, Federal District
  - Hospital de Messejana Dr. Carlos Alberto Studart Gomes, Goiânia, Goiás
  - Hospital Ruy Azeredo, Goiânia, Goiás
  - Instituto Goiano de Oncologia e Hematologia - INGOH, Goiânia, Goiás
  - Hospital Felicio Rocho, Belo Horizonte, Minas Gerais
  - NUPEC-Orizonti, Belo Horizonte, Minas Gerais
  - Hospital Santa Cruz, Curitiba, Paraná
  - PUCPR, Curitiba, Paraná
  - Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - Hospital Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Universitario de Santa Maria, Santa Maria, Rio Grande do Sul
  - Hospital Sao Jose, Criciúma, Santa Catarina
  - Hospital Regional Homero Miranda Gomes, São José, South Carolina
  - Hospital de Reabilitacao de Anomalias Craniofaciais, Bauru, São Paulo
  - UPECLIN - Unidade de Pesquisa Clínica da Faculdade de Medicina de Botucatu, Botucatu, São Paulo
  - Hospital Universitario Sao Francisco na Providencia na Deus, Bragança Paulista, São Paulo
  - Fundação Centro Médico de Campinas, Campinas, São Paulo
  - IPECC, Campinas, São Paulo
  - CiTen - Centro Hospital Municipal Antonio Giglio, Osasco, São Paulo
  - Hospital Regional de Presidente Prudente, Presidente Prudente, São Paulo
  - Hospital Estadual de Serrana, Ribeirão Preto, São Paulo
  - HCFMUSP, São Paulo, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo
  - Santa Casa de Misericordia de Sao Paulo, São Paulo, São Paulo
- Canada (25):
  - Foothills Medical Centre, Calgary, Alberta
  - Grand Prairie Regional Hospital, Grande Prairie, Alberta
  - Nanaimo Regional General Hospital, Nanaimo, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Health Sciences Center Winnipeg, Winnipeg, Manitoba
  - Grace General Hospital, Winnipeg, Manitoba
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Memorial University, St. John's, Newfoundland and Labrador
  - Health Sciences North Research Institute, Greater Sudbury, Ontario
  - Hamilton Health Sciences - Juravinski, Hamilton, Ontario
  - Hamilton Health Sciences, Hamilton, Ontario
  - Markham Stouffville Hospital, Markham, Ontario
  - Hôpital Montfort, Ottawa, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Niagara Health System - St Catharines Site, Saint Catherines, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Centre Hospitalier de Quebec - Hotel-Dieu de Levis, Lévis, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Centre Hospitalier de l'université de Montréal (CHUM), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec-University Laval, Québec, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec (IUCPQ), Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Regina General Hospital, Regina, Saskatchewan

REFERENCES:
- [Background] ATTACC Investigators; ACTIV-4a Investigators; REMAP-CAP Investigators; Lawler PR, Goligher EC, Berger JS, Neal MD, McVerry BJ, Nicolau JC, Gong MN, Carrier M, Rosenson RS, Reynolds HR, Turgeon AF, Escobedo J, Huang DT, Bradbury CA, Houston BL, Kornblith LZ, Kumar A, Kahn SR, Cushman M, McQuilten Z, Slutsky AS, Kim KS, Gordon AC, Kirwan BA, Brooks MM, Higgins AM, Lewis RJ, Lorenzi E, Berry SM, Berry LR, Aday AW, Al-Beidh F, Annane D, Arabi YM, Aryal D, Baumann Kreuziger L, Beane A, Bhimani Z, Bihari S, Billett HH, Bond L, Bonten M, Brunkhorst F, Buxton M, Buzgau A, Castellucci LA, Chekuri S, Chen JT, Cheng AC, Chkhikvadze T, Coiffard B, Costantini TW, de Brouwer S, Derde LPG, Detry MA, Duggal A, Dzavik V, Effron MB, Estcourt LJ, Everett BM, Fergusson DA, Fitzgerald M, Fowler RA, Galanaud JP, Galen BT, Gandotra S, Garcia-Madrona S, Girard TD, Godoy LC, Goodman AL, Goossens H, Green C, Greenstein YY, Gross PL, Hamburg NM, Haniffa R, Hanna G, Hanna N, Hegde SM, Hendrickson CM, Hite RD, Hindenburg AA, Hope AA, Horowitz JM, Horvat CM, Hudock K, Hunt BJ, Husain M, Hyzy RC, Iyer VN, Jacobson JR, Jayakumar D, Keller NM, Khan A, Kim Y, Kindzelski AL, King AJ, Knudson MM, Kornblith AE, Krishnan V, Kutcher ME, Laffan MA, Lamontagne F, Le Gal G, Leeper CM, Leifer ES, Lim G, Lima FG, Linstrum K, Litton E, Lopez-Sendon J, Lopez-Sendon Moreno JL, Lother SA, Malhotra S, Marcos M, Saud Marinez A, Marshall JC, Marten N, Matthay MA, McAuley DF, McDonald EG, McGlothlin A, McGuinness SP, Middeldorp S, Montgomery SK, Moore SC, Morillo Guerrero R, Mouncey PR, Murthy S, Nair GB, Nair R, Nichol AD, Nunez-Garcia B, Pandey A, Park PK, Parke RL, Parker JC, Parnia S, Paul JD, Perez Gonzalez YS, Pompilio M, Prekker ME, Quigley JG, Rost NS, Rowan K, Santos FO, Santos M, Olombrada Santos M, Satterwhite L, Saunders CT, Schutgens REG, Seymour CW, Siegal DM, Silva DG Jr, Shankar-Hari M, Sheehan JP, Singhal AB, Solvason D, Stanworth SJ, Tritschler T, Turner AM, van Bentum-Puijk W, van de Veerdonk FL, van Diepen S, Vazquez-Grande G, Wahid L, Wareham V, Wells BJ, Widmer RJ, Wilson JG, Yuriditsky E, Zampieri FG, Angus DC, McArthur CJ, Webb SA, Farkouh ME, Hochman JS, Zarychanski R. Therapeutic Anticoagulation with Heparin in Noncritically Ill Patients with Covid-19. N Engl J Med. 2021 Aug 26;385(9):790-802. doi: 10.1056/NEJMoa2105911. Epub 2021 Aug 4. PMID 34351721